CLINICAL TRIAL: NCT04055493
Title: Adjuvant Dynamic Marker - Adjusted Personalized Therapy Comparing Endocrine Therapy Plus Ribociclib Versus Chemotherapy in Intermediate Risk, HR+/HER2- Early Breast Cancer
Brief Title: Adj. Marker-adjusted Personalized Therapy Comparing ET+Ribociclib vs Chemotherapy in Intermediate Risk, HR+/HER2- EBC
Acronym: ADAPTcycle
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Novartis (Industry); Genomic Health®, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM08 (ADAPTcycle)
Record Dates: First submitted 2019-07-22; First posted 2019-08-13 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Female
Keywords: early breast cancer; ADAPT; endocrine therapy; ribociclib; intermediate risk; HER2 negative; HR positive
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Tablets

STUDY DESIGN:
Intervention Model Description: Multicenter, interventional, prospective, two-arm, randomized, open-label, controlled (neo)adjuvant, phase-III trial evaluating the efficacy and safety of ribociclib combined with endocrine therapy (ET) versus standard-of-care chemotherapy in early breast cancer (EBC) patients with molecular HR+/HER2- subtype.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ribociclib plus ET (Experimental): Ribociclib 600mg / day over 26 cycles + endocrine treatment of physician´s choice
  Interventions: Drug: Ribociclib 200Mg Oral Tablet
- Standard-of-care chemotherapy (No Intervention): Standard-of-care chemotherapy according to the clinical guidelines, e.g., of the Breast Committee of the German Gynecological Oncology Group (AGO), and regional prescribing information depending on patient's needs for 16-24 weeks,

INTERVENTIONS:
Drug: Ribociclib 200Mg Oral Tablet — 3 x 200 MG per os
  Other Names: Kisqali
  Arms: Ribociclib plus ET

SUMMARY:
The study investigates, whether the patient group with intermediate-risk early breast cancer benefits from treatment with ribociclib in combination with endocrine therapy compared to standard-of-care chemotherapy (followed by adjuvant endocrine therapy).

DETAILED DESCRIPTION:
The WSG ADAPT trial program is one of the first new generation trials addressing the issue of individualization of (neo)-adjuvant decision-making in early breast cancer (EBC) in a subtype-specific manner. The first WSG ADAPT umbrella trial (NCT01779206) aimed to establish early predictive molecular surrogate markers for response after a short 3-week induction treatment.

The goals of the WSG ADAPT trial program - early response assessment and subtype-specific therapy tailoring to those patients who are most likely to benefit - have contributed to the very positive national and international feedback to the ADAPT concept as a whole.

The aim of this ADAPTcycle phase-III-trial is to investigate whether the intermediate-risk patient group identified during the screening phase derives additional benefit from treatment with ribociclib in combination with ET compared to chemotherapy (followed by adjuvant ET).

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

A. Prior to REGISTRATION in the study:

1. Written informed consent prior to any screening procedures. 2. Female. 3. ≥ 18 years of age. 4a. EITHER: (Post)menopausal status at the time of initiation of (neo)adjuvant study medication

* patient underwent bilateral oophorectomy, or
* age ≥ 60, or
* age < 60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) and/or FSH and estradiol in the postmenopausal range per local normal range.

  4b. OR: Pre-menopausal patients:
* confirmed negative serum pregnancy test (β-hCG) before starting study treatment, or
* patient has had a hysterectomy. 5. Histologically confirmed diagnosis of primary estrogen-receptor positive and/or progesterone-receptor positive (> 1%) early breast cancer by local laboratory.

  6. Patient has HER2-negative breast cancer defined as
* a negative in-situ hybridization test or an IHC status of 0, 1+, or 2+,
* if IHC is 2+, a negative in-situ hybridization (FISH, CISH, or SISH) test is required (based on the most recently analyzed tissue sample and all tested by a local laboratory).

  7. Local therapy of breast cancer (if adjuvant treatment or planned if neoadjuvant treatment) according to current guidelines.

Note: This may include radiotherapy of breast cancer.

B. Prior to RANDOMIZATION in the study 8. No evidence of distant metastasis (confirmed prior to randomization by, preferentially, CT thorax / abdomen, X-ray chest, ultrasound liver, bone scan, or PET-CT).

9. Patient has available tumor tissue from diagnostic biopsy. 10. Patient is classified as intermediate risk according to the ADAPT intermediate-risk definition (i) (as follows), or (only in case of missing Oncotype DX or Ki-67 response data), according to the clinical intermediate-risk definition (ii) (as follows).

(i). ADAPT intermediate-risk definition: Patient meets one of the following criteria:

* c/pN0, RS ≤ 25 with luminal-B-like (Ki-67 ≥20% or G3) or c/pT2-4 without endocrine response (post-endocrine Ki-67 > 10 %)
* c/pN1, RS ≤ 25 without endocrine response (post-endocrine Ki-67 > 10 %)
* c/pN0, RS > 25 with luminal-B-like (Ki-67 ≥20% or G3) or c/pT2-4 with endocrine response (Ki-67 ≤ 10 %)
* c/pN1, RS > 25 with endocrine response (Ki-67 ≤ 10 %)
* c/pN2-3, RS ≤ 25 with endocrine response (Ki-67 ≤ 10 %). Note: Postmenopausal patients with pT1-2/pN0 disease and RS < 25, as well as premenopausal patients with pT1-2/pN0 disease and RS<16, are recommended to be treated by endocrine therapy alone and not to be randomized (at investigator´s discretion).

(ii). Clinical intermediate-risk definition (ascertained by investigator): Clinical intermediate risk may be ascertained by the investigator prior to randomization if at maximum two of the following three risk factors are present (according to primary diagnosis / 1st sample):

1. cT2-4
2. c/pN positive
3. G3 and / or Ki-67 ≥ 20% Note: Inclusion of a patient according to "clinical intermediate risk" is permitted only in case of missing baseline Oncotype DX® or Ki-67 decrease. In this case, investigators will follow a risk-based, step-wise assessment process.

11. No contraindication for (neo)-adjuvant ET. 12. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1. 13. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

* absolute neutrophil count ≥ 1.5 × 109/L,
* platelets ≥ 100 × 109/L,
* hemoglobin ≥ 9.0 g/dL,
* estimated glomerular filtration rate (eGFR) ≥ 30 mL/min by a Cockcroft-Gault formula,
* INR ≤ 1.5,
* serum creatinine < 1.5 mg/dL,
* total bilirubin < ULN, except for patients with Gilbert's Syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN,
* aspartate transaminase (AST) < 2.5 × ULN,
* alanine transaminase (ALT) < 2.5 × ULN. 14. 2-lead-ECG (CANKADO) with:
* QTcF interval at screening < 450 msec (using Fridericia's correction),
* mean resting heart rate 50-90 bpm (determined from the ECG). 15. Ability to swallow ribociclib tablets or to administer other study medication, respectively.

  16. Ability to communicate with the investigator and comply with study procedures.

  17. Willing to remain during therapy at the clinical site, as required by the protocol.

Exclusion Criteria:

Patients eligible for inclusion in this study must not meet any of the following criteria:

1. Patient with distant metastases of breast cancer beyond regional lymph nodes.
2. Patient has received prior (neo)-adjuvant treatment with chemotherapy, ET, or any CDK4/6 inhibitor for breast cancer.
3. Patient has received tamoxifen, raloxifene, or aromatase inhibitors (AIs) for reduction in risk ("chemoprevention") of breast cancer and/or treatment for osteoporosis within last 2 years prior to screening.
4. Patient has received prior neoadjuvant/adjuvant treatment with anthracyclines at cumulative doses of 450 mg/m² or more for doxorubicin or 900 mg/m² or more for epirubicin.
5. Patient with a known hypersensitivity to any of the excipients of ribociclib, ET, or standard-of-care chemotherapy.
6. Patient with inflammatory breast cancer at screening.
7. Patient is concurrently using other anti-cancer therapy.
8. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects.
9. Patient is currently receiving warfarin or other coumarin-derived anti-coagulant for treatment, prophylaxis, or otherwise.
10. Patient has not recovered from clinical and laboratory acute toxicities related to prior anticancer therapies to NCI CTCAE version 5.0 Grade ≤ 1.
11. Patient has a concurrent malignancy, or malignancy within 5 years of randomization, or known history of invasive breast cancer.
12. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small-bowel resection).
13. Patient has a known history of HIV infection.
14. Patient has known active hepatitis-B-virus (HBV) or hepatitis-C-virus (HCV) infection.
15. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator´s judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study, or compromise compliance with the protocol (e.g., chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial, or viral infections, etc.).
16. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

    * history of myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry,
    * documented cardiomyopathy,
    * left ventricular ejection fraction (LVEF) < 50 % as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO),
    * long QT syndrome, family history of idiopathic sudden death, congenital long QT syndrome, or any of the following:

      * risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/ symptomatic bradycardia,
      * concomitant medications with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g., within 5 half-lives or 7 days prior to starting study drug),
      * inability to determine the QTcF interval,
      * clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left-bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II, and 3rd-degree AV block),
      * systolic blood pressure (SBP) > 160 or < 90 mmHg.
17. Patient is currently receiving any of the following substances, which cannot be discontinued 7 days prior to Cycle 1 Day 1:

    * concomitant medications, herbal supplements, fruits (e.g. grapefruit, pomegranates, pomelos, star fruit, Seville oranges) and their juices that are strong inducers or inhibitors of CYP3A4/5,
    * medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
18. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.
19. Participation in a prior investigational study within 30 days prior to enrollment or within five half-lives of the investigational product, whichever is longer.
20. Not able to understand and to comply with study instructions and requirements.
21. Pregnant or nursing (lactating) woman.
22. Woman of child-bearing potential defined as woman physiologically capable of becoming pregnant, unless she is using highly effective methods of contraception during the study treatment and for 21 days after stopping the treatment:

    * total abstinence (when this is in line with the preferred and usual lifestyle of the patient).
    * female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment.
    * male partner sterilization (at least 6 months prior to study screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient.
    * placement of an intrauterine device (IUD).
23. Use of oral (estrogen and progesterone), transdermal, injected, or implanted hormonal methods of contraception as well as hormonal replacement therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pre- and postmenopausal women 18 years or older.
Enrollment: 1684 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
invasive disease-free survival (iDFS) | at end of study, on average 5 years after start of treatment
  superiority in invasive disease-free survival (iDFS) of ribociclib + ET vs. standard-of-care chemotherapy
distant disease-free survival (dDFS) | at end of study, on average 5 years after start of treatment
  distant disease-free survival (dDFS) in the ribociclib + ET-group to demonstrate survival rate >92%

SECONDARY OUTCOMES:
overall survival (OS) 95 % CI | at end of study, on average 5 years after start of treatment
  95 %-confidence interval (CI) for OS in both arms
distant disease-free survival (dDFS) 95 % CI | at end of study, on average 5 years after start of treatment
  95 %-confidence interval (CI) for dDFS in both arms
QoL | at end of study, on average 5 years after start of treatment
  quality of life (QoL) and correlation to treatment-related symptoms measured by EQ-VAS and triggered symptom questionnaire,
treatment adherence | at end of study, on average 5 years after start of treatment
  treatment adherence measured by drug intake compared between treatment arms
pathological complete response (pCR) | at end of study, on average 5 years after start of treatment
  Pathological response rate (defined as ypT0/is/ypN0), as well as further definitions (ypT0/ypN0; ypT0/is/any ypN, near pCR (ypT1a/any ypN)), in neoadjuvant treated patients
clinical response rate | at end of study, on average 5 years after start of treatment
  clinical response rate (by palpation, ultrasound, and further methods) compared between treatment arms
rate of breast-conservation therapy | at end of study, on average 5 years after start of treatment
  prevalence of breast conservation therapy vs. mastectomy compared between treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr., Principal Investigator — Ludwigs-Maximilians-University Munich, Breast Cancer Centre
Locations (86):
- Germany (86):
  - Ost-Alb Klinikum Brustzentrum, Aalen, Baden-Wurttemberg
  - Stadtklinik Baden-Baden Brustzentrum, Baden-Baden, Baden-Wurttemberg
  - Kreiskliniken Böblingen Klinikum Böblingen Frauenklinik, Böblingen, Baden-Wurttemberg
  - Uniklinikum Freiburg Frauenklinik, Freiburg im Breisgau, Baden-Wurttemberg
  - Praxis für interdisziplinäre Onkologie & Hämatologie GbR Praxis am Diakonieklinikum, Freiburg im Breisgau, Baden-Wurttemberg
  - SLK-Kliniken-Heilbronn Frauenklinik, Heilbronn, Baden-Wurttemberg
  - Klinikum Ludwigsburg Klinik für Frauenheilkunde u. Geburtshilfe, Ludwigsburg, Baden-Wurttemberg
  - Universitätsklinikum Tübingen Universitäts-Frauenklinik, Tübingen, Baden-Wurttemberg
  - Universitätsfrauenklinik Ulm Frauenheilkunde und Geburtshilfe, Ulm, Baden-Wurttemberg
  - GRN Klinik Weinheim Gynäkologie, Weinheim, Baden-Wurttemberg
  - Klinikum der Universität München Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Brustzentrum, Munich, Bavaria
  - Rotkreuzkliniken München Frauenklinik - Gynäkologie, München, Bavaria
  - Frauenklinik und Poliklinik / Studienzentrale Josef-Schneider-Straße 4, Würzburg, Bavaria
  - Carl-Thiem-Klinikum / Brustzentrum Senologie der Frauenklinik, Cottbus, Brandenburg
  - Schwerpunktpraxis Gynäkologische Onkologie Praxis Dr. Heinrich, Fürstenwalde, Brandenburg
  - Klinikum Ernst von Bergmann Klinik für Gynäkologie und Geburtshilfe, Potsdam, Brandenburg
  - Klinikum Bremerhaven Reinkenheide Frauenklinik, Bremerhaven, City state Bremen
  - AGAPLESION Markus Krankenhaus / Brustzentrum Gynäkologie und Geburtshilfe, Frankfurt am Main, Hesse
  - Klinikum Frankfurt Höchst Klinik für Gynäkologie und Geburtshilfe, Frankfurt am Main, Hesse
  - Klinikum Kassel Frauenklinik, Kassel, Hesse
  - Sana Klinikum Klinik für Gynäkologie und Geburtshilfe, Studienambulanz AOZ, Offenbach, Hesse
  - St. Josefs-Hospital Wiesbaden Frauenklinik - Gynäkologie, Wiesbaden, Hesse
  - Frauenärzte Casparistraße Studien GbR BS, Braunschweig, Lower Saxony
  - MVZ II der Niels Stensen Kliniken Onkologie u. Hämatologie, Brustzenzrum, Georgsmarienhütte, Lower Saxony
  - Medizinische Hochschulle Hannover Klinik für Frauenheilkunde und Geburtshilfe, Hanover, Lower Saxony
  - DIAKOVERE Henriettenstift Frauenklinik, Hanover, Lower Saxony
  - Gynäkologische Gemeinschaftspraxis-Ärztehaus am Bahnhofsplatz Klinische Studien, Hildesheim, Lower Saxony
  - Städtisches Klinikum Lüneburg Frauenklinik, Lüneburg, Lower Saxony
  - MVZ Klinik Dr. Hancken Haematologie/Onkologie, Stade, Lower Saxony
  - UFK Klinikum Südstadt Frauenklinik, Rostock, Mecklenburg-Vorpommern
  - Marienhospital Studienzentrale BrustCentrum Aachen-Kreis Heinsberg, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Aachen, Frauenklinik - Senologie, Aachen, North Rhine-Westphalia
  - EVK Bergisch Gladbach Brustzentrum, Bergisch Gladbach, North Rhine-Westphalia
  - Onkologische Schwerpunktpraxis Bielefeld Praxis Dr. Just, Bielefeld, North Rhine-Westphalia
  - Marienhospital Bottrop Klinik für Gynäkologie und Geburtshilfe / Gyn-Ambulanz, Bottrop, North Rhine-Westphalia
  - St. Elisabeth-Krankenhaus Hohenlind Brustzentrum, Cologne, North Rhine-Westphalia
  - Uniklinik Köln / Gebäude 70 Studienzentrale der Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Cologne, North Rhine-Westphalia
  - Kliniken der Stadt Köln / Krankenhaus Holweide Brustzentrum Holweide, Cologne, North Rhine-Westphalia
  - Klinikum Dortmund gGmbH Frauenklinik, Dortmund, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf Klinik für Frauenheilkunde & Geburtshilfe, Düsseldorf, North Rhine-Westphalia
  - Luisenkrankenhaus GmbH GynOnco Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Praxis Dr. Adhami, Erkelenz, North Rhine-Westphalia
  - St. Antonius Hospital Klinik für Hämatologie/Onkologie, Eschweiler, North Rhine-Westphalia
  - Universitätsklinikum Essen Klinik für Frauenheilkunde und Geburtshilfe, Essen, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Klinik für Senologie/Interdisziplinäres Brustzentrum, Essen, North Rhine-Westphalia
  - Evangelische Kliniken Gelsenkirchen GmbH Klinik für Senologie, Gelsenkirchen, North Rhine-Westphalia
  - Wilhelm-Anton-Hospital Goch Klinik für Innere Medizin, Hämatologie u. Onkologie, Goch, North Rhine-Westphalia
  - Onkodok GmbH, Gütersloh, North Rhine-Westphalia
  - St. Barbara Klinik Brustzentrum, Hamm, North Rhine-Westphalia
  - Klinikum Leverkusen Medizinische Klinik 3, Leverkusen, North Rhine-Westphalia
  - Praxis für gynäkologische Onkologie am Ev. Krankenhaus Bethesda, Mönchengladbach, North Rhine-Westphalia
  - St. Franziskus-Hospital Brustzentrum, Münster, North Rhine-Westphalia
  - Universitätsklinikum Frauenheilkunde, Münster, North Rhine-Westphalia
  - ONCOLOGIANOVA Praxis Dr. Emde, Recklinghausen, North Rhine-Westphalia
  - Marienkrankenhaus Schwerte Brustzentrum, Schwerte, North Rhine-Westphalia
  - Marien-Krankenhaus Klinik für Gynäkologie und Geburtshilfe, Siegen, North Rhine-Westphalia
  - Diakonie Klinikum Jung Stilling Brustzentrum, Siegen, North Rhine-Westphalia
  - Praxisnetz Hämatologie / internistische Onkologie Praxis Troisdorf, Troisdorf, North Rhine-Westphalia
  - Christliches Klinikum Unna gGmbH Brustzentrum, Unna, North Rhine-Westphalia
  - Praxis für Hämatologie und internistische Onkologie Praxis Dr. Nusch, Velbert, North Rhine-Westphalia
  - Marien Hospital / Senologie Brustzentrum, Witten, North Rhine-Westphalia
  - Helios Universitätsklinikum Frauenheilkunde & Geburtshilfe, Wuppertal, North Rhine-Westphalia
  - Katholisches Klinikum Koblenz-Montabaur-Marienhof Koblenz Marienhof Koblenz - Gynäkologie, Koblenz, Rhineland-Palatinate
  - Klinikum Mutterhaus der Borromäerinnen Innere Medizin I / Onkologie, Trier, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes Frauenklinik, Homburg, Saarland
  - DRK Kliniken Saar / Krankenhaus Saarlouis Brustzentrum, Saarlouis, Saarland
  - Klinikum Chemnitz Frauenklinik / Brustzentrum, Chemnitz, Saxony
  - Universitätsklinikum Dresden Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Dresden, Saxony
  - Universitätsklinikum Leipzig Gynäkologie und Universitäres Krebszentrum; Klinik und Poliklinik für Frauenheilkunde, Leipzig, Saxony
  - Kliniken St. Georg Klinik für Gynäkologie und Geburtshilfe, Leipzig, Saxony
  - Klinikum Obergöltzsch-Rodewisch Frauenklinik, Rodewisch, Saxony
  - Universitätsklinikum Halle Universitätsklinik für Gynäkologie, Halle, Saxony-Anhalt
  - Altmark-Klinikum Salzwedel Klinik für Frauenheilkunde, Salzwedel, Saxony-Anhalt
  - Johanniter Frauenklinik Stendal Gynäkologie, Stendal, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Frauenklinik, Lübeck, Schleswig-Holstein
  - Universitätsklinikum Jena Klinik und Poliklinik für Frauenheilkunde und Fortpflanzungsmedizin, Jena, Thuringia
  - MVZ Nordhausen Praxis Dr. Andrea Grafe, Nordhausen, Thuringia
  - Charité Berlin, Klinik für Gynäkologie m.S. Senologie Brustzentrum (CCM), Berlin
  - St. Gertrauden Krankenhaus Brustzentrum City Berlin, Berlin
  - Vivantes Klinikum Am Urban Brustzentrum, Berlin
  - DRK Klinikum Berlin-Köpenick Brustzentrum, Berlin
  - Evangelisches Waldkrankenhaus Spandau Klinik für Gynäkologie und Geburtshilfe, Berlin
  - Hämatologisch/Onkologische Schwerpunktpraxis Praxis Dr. Schreiber, Bremen
  - UKE Hamburg / Frauenklinik Brustzentrum am UKE, Hamburg
  - Agaplesion Diakonieklinikum Hamburg Frauenklinik, Brustzentrum u. Gyn. Tumorzentrum / Gyn. Studienambulanz, Hamburg
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
The sponsor is committed to following high ethical standards for reporting study results, including the timely communication and publication of clinical trial results, whatever their outcome. The sponsor assures that the key design elements of this protocol will be posted on a publicly accessible database, e.g., www.clinicaltrials.gov, before study start.
  As part of its commitment to full transparency in publications, the sponsor supports the full disclosure of all funding sources for the study and publications, as well as any actual and potential conflicts of interest of financial and non-financial nature by all authors, including medical writing / editorial support, if applicable.
Supporting Information: CSR
Time Frame: Within 1 year after end of study.
Access Criteria: for regulatory use only

REFERENCES:
- [Derived] Klier K, Patel YJ, Schinkothe T, Harbeck N, Schmidt A. Corrected QT Interval (QTc) Diagnostic App for the Oncological Routine: Development Study. JMIR Cardio. 2023 Sep 11;7:e48096. doi: 10.2196/48096. PMID 37695655